CLINICAL TRIAL: NCT04931316
Title: Incidence and Management of Ocular Hypertension Following Deep Anterior Lamellar Keratoplasty
Acronym: Dalk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amgad Mahmoud El Nokrashy, Lecturer of Ophthalmology, Mansoura University
Other Study IDs: R.20.12.1121
Record Dates: First submitted 2021-06-12; First posted 2021-06-18 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Unrecognized Condition
MeSH Terms: interventions — Antiglaucoma Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: antiglaucoma — use antiglaucoma in ocular hypertension

SUMMARY:
This is a retrospective case series study that included patients who performed deep anterior lamellar keratoplasty and presented with elevated intraocular pressure during follow up.

DETAILED DESCRIPTION:
This is a retrospective case series study that included patients who performed deep anterior lamellar keratoplasty and presented with elevated intraocular pressure during follow up. Patients' demographic characteristics, medical, and ocular history will be recorded.

Inclusion criteria will include patients who were diagnosed with elevated intraocular pressure (IOP) after DALK surgery performed from 2018 to 2020 with follow up duration more than 6 months. Patients with less than 6 months of follow-up will be excluded from the study.

Patients' demographic characteristics, medical and ocular history will be recorded. Baseline complete ophthalmic examination was performed. It included best corrected visual acuity (BCVA) using Landolt C chart that was converted to log minimum angle of resolution (log MAR) for statistical analysis, slit lamp anterior segment examination (with attention to cornea, bulbar conjunctiva and AC), intraocular pressure measurement using rebound system (I care tonometer, Topcon, Canada), angle assessment and fundus examination using Goldman 3 mirror contact lens.

High IOP was defined as intraocular pressure more than 25 mmHg. Data will be collected with attention to appropriate management done either medical treatment or surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed with elevated IOP after DALK surgery performed from 2018 to 2020

Exclusion Criteria:

* Patients with penetrating keratoplasty

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with DALK
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure values | this is a retrospective study . collection of data from patients records over 2 months
  assessment of intraocular pressure after lamellar keratoplasty

CONTACTS AND LOCATIONS:
Overall Officials: AHMED El WEHEDY, MD, Principal Investigator — Mansoura University; Hatem El Awady, MD, Study Chair — Mansoura University; AYA HASHISH, MD, Study Chair — Mansoura University; AMGAD EL NOKRASHY, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No